CLINICAL TRIAL: NCT04269057
Title: Change of NLRP3 Inflammasome Expression Level, Symptoms, and Functional Status in Patients With Heart Failure With Preserved Ejection Fraction Treated With ARNI
Brief Title: Change of NLRP3 Inflammasome Expression Level, Symptoms, and Functional Status in HFpEF Patients Treated With ARNI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Associate Professor, Chongqing Medical University
Other Study IDs: 2019-10
Record Dates: First submitted 2020-01-13; First posted 2020-02-13 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure
Keywords: NLRP3 protein; human
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — monocytes and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HFpEF: heart failure patients with preserved ejection fraction who using ARNI
- HFrEF: heart failure patients with reduced ejection fraction who using ARNI

SUMMARY:
Underlying inflammation has been increasingly recognized in heart failure with a preserved ejection fraction(HFpEF). But there is no study reported the relationship between NLRP3 inflammasome and HFpEF. In this study, investigators propose a scientific hypothesis that the expression of NLRP3 inflammasome is elevated in patients with HFpEF, and the level of TNFα, IL-1β and NLRP3 inflammasome is lower in patients treated with sacubitril/valsartan.

DETAILED DESCRIPTION:
The study will integrate data from two trials involving a total of 90 participants with heart failure. Depending on the using of ARNI, participants in HFpEF group will be divided into two groups. The diagnostic criteria for HFpEF is: (1) left ventricular ejection fraction ≥50%； (2）with the symptoms and/or signs of heart failure; (3) BNP≥35 pg/mL and/or NTproBNP≥125 pg/mL; (4) at least one additional criterion: a.relevant structural heart disease(LVH and/or LAE); b.diastolic dysfunction. The primary outcome are the change from baseline in TNFα, IL-1β, NLRP3 inflammasome, and so on assessed at 12 weeks. The key secondary outcomes include changes in echocardiographic measures, quality of life, etc. And then compare the rate of above indicators of two trials.

ELIGIBILITY:
Inclusion Criteria:

* left ventricular ejection fraction ≥50%；
* with the symptoms and/or signs of heart failure；
* BNP≥35 pg/mL and/or NTproBNP≥125 pg/mL；
* at least one additional criterion: relevant structural heart disease(LVH and/or LAE) or diastolic dysfunction.

Exclusion Criteria:

* LVEF less than 45% at any time;
* severe infection;
* ACS;
* pregnancy;
* eGFR <30 mL/min/1.73 m2, etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: heart failure patients
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in TNFα, IL-1β, NLRP3 inflammasome, and so on assessed at 12 weeks | 12 weeks
  Measuring the level of TNFα, IL-1β, NLRP3 inflammasome, and so on from blood samples at 12 weeks, seperately by PCR and ELISA

SECONDARY OUTCOMES:
The change from baseline in echocardiographic measures and so on | 12 months
  Observed the change of ejection fraction, left atrial volume index and so on measured by echocardiogram.
The change from baseline in quality of life | 12 months
  Measured by Kansas City Cardiomyopathy Questionnaire. The score ranges from 0 to 100. The higher score means the better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, doctor, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China